CLINICAL TRIAL: NCT05513703
Title: Phase 2, Open-Label Study in Subjects With Previously Untreated MET Amplified Locally Advanced/Metastatic Non-Squamous Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study to Assess Disease Activity of Intravenously (IV) Infused Telisotuzumab Vedotin in Adult Participants With Advanced/Metastatic Non-Squamous Non-Small Cell Lung Cancer (NSCLC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic considerations
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M22-137; 2022-500608-23-00 (Other: EU CT)
Expanded Access: NCT04830202 (Available)
Record Dates: First submitted 2022-08-23; First posted 2022-08-24 (Actual); Results first posted 2025-10-24 (Actual); Last update posted 2025-10-24 (Actual); Status verified 2025-10

CONDITIONS: Non Small Cell Lung Cancer
Keywords: c-Met NSCLC; Telisotuzumab Vedotin; ABBV-399; Cancer; Non Small Cell Lung Cancer; NSCLC; MET Amplified NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — telisotuzumab vedotin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Telisotuzumab Vedotin (Experimental): Participants will receive telisotuzumab vedotin every 2 weeks until meeting study drug discontinuation criteria.
  Interventions: Biological: Telisotuzumab Vedotin

INTERVENTIONS:
Biological: Telisotuzumab Vedotin — Intravenous (IV) Infusion
  Other Names: ABBV-399

SUMMARY:
Cancer is a condition where cells in a specific part of body grow and reproduce uncontrollably. Non-small cell lung cancer (NSCLC) is a solid tumor, a disease in which cancer cells form in the tissues of the lung. The purpose of this study is to determine how telisotuzumab vedotin affects the disease state in adult participants with previously untreated participants with MET amplified non-squamous NSCLC. Change in disease activity will be assessed.

Telisotuzumab vedotin is an investigational drug being developed for the treatment of MET amplified non-squamous NSCLC. Participants receive intravenously (IV) infused of telisotuzumab vedotin. Approximately 70 adult participants with previously untreated MET amplified locally advanced/metastatic non-squamous NSCLC will be enrolled in the study in approximately 110 sites worldwide.

Participants will receive IV telisotuzumab vedotin every 2 weeks until meeting study drug discontinuation criteria.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at a hospital or clinic. The effect of the treatment will be checked by medical assessments, blood tests, checking for side effects and completing questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Must have MET amplification in tumor tissue as determined by the Sponsor-designated central laboratory MET FISH Assay or in plasma and/or tissue by a Sponsor-approved assay.
* Must have histologically documented non-squamous adenocarcinoma non-small cell lung cancer (NSCLC) that is locally advanced or metastatic.
* Must have measurable disease per Response Evaluation Criteria in Solid Tumors (RECIST) version 1.1.
* Must have an Eastern Cooperative Oncology Group (ECOG) Performance Status of 0 or 1.
* Participant may have received prior adjuvant/neoadjuvant systemic chemotherapy and/or radiation and/or immunotherapy provided that the subject has not progressed on or within 6 months of completing the regimen and it was completed >= 6 months before subject's first dose of study drug.
* Metastases to the central nervous system (CNS) are eligible only after definitive therapy is provided as noted in the protocol.
* History of radiation pneumonitis in the radiation field (fibrosis) is permitted.

Exclusion Criteria:

* Alterations in EGFR, ALK, ROS1, or BRAF that predict sensitivity to available targeted therapy. Participants with other alterations that are candidates for available targeted therapy.
* Prior systemic therapy for locally advanced/metastatic NSCLC. Of note, limited treatment with no more than 1 cycle of chemotherapy is allowed prior to receiving the first dose of study drug provided there is no evidence of progression.
* Have a history of other malignancies except those noted in the protocol.
* Have a history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan.
* Received prior c-Met-targeted antibodies.
* Have NSCLC that is eligible for treatment with curative intent.
* Have unresolved adverse events (AEs) >= Grade 2 from prior anticancer therapy, except for alopecia or anemia.
* Have had major surgery within 21 days prior to the first dose of telisotuzumab vedotin.
* Have clinically significant condition(s) as noted in the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-11-21 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (29):
- United States (2):
  - Cancer and Blood Speciality Clinic - Los Alamitos /ID# 251671, Los Alamitos, California
  - Valley Medical Center /ID# 251880, Renton, Washington
- Monash Health - Monash Medical Centre /ID# 247679, Clayton, Victoria, Australia
- France (3):
  - CHU Lille - Hôpital Albert Calmette /ID# 246263, Lille, Hauts-de-France
  - Hospices Civils de Lyon (HCL) - Hopital Louis Pradel /ID# 246267, Bron, Rhone
  - Centre Jean Perrin /ID# 246268, Clermont-Ferrand
- Asklepios Fachkliniken Muenchen-Gauting /ID# 248082, Gauting, Germany
- Israel (5):
  - Meir Medical Center /ID# 243208, Kfar Saba, Central District
  - Rambam Health Care Campus /ID# 246781, Haifa, H_efa
  - Hadassah Medical Center-Hebrew University /ID# 243298, Jerusalem, Jerusalem
  - The Chaim Sheba Medical Center /ID# 243207, Ramat Gan, Tel Aviv
  - Rabin Medical Center /ID# 248631, Petah Tikva
- Italy (3):
  - Duplicate_Fondazione IRCCS San Gerardo dei Tintori /ID# 247584, Monza, Monza E Brianza
  - Istituto di Candiolo Fondazione del Piemonte per l'Oncologia IRCCS /ID# 248329, Candiolo, Torino
  - IRCCS Istituti Fisioterapici Ospitalieri-Istituto Nazionale Tumori Regina Elena /ID# 247585, Rome
- Japan (6):
  - National Cancer Center Hospital East /ID# 250317, Kashiwa-shi, Chiba
  - Duplicate_National Hospital Organization Kyushu Cancer Center /ID# 250714, Fukuoka, Fukuoka
  - Hokkaido University Hospital /ID# 250316, Sapporo, Hokkaido
  - Osaka International Cancer Institute /ID# 251507, Osaka, Osaka
  - Shizuoka Cancer Center /ID# 251752, Sunto-gun, Shizuoka
  - National Cancer Center Hospital /ID# 250319, Chuo-ku, Tokyo
- South Korea (4):
  - Keimyung University Dongsan Hospital /ID# 247371, Daegu, Gyeongsangbuk-do
  - Pusan National University Yangsan Hospital /ID# 248489, Yangsan, Gyeongsangnam-do
  - Chungbuk National University Hospital /ID# 248405, Cheongju-si, North Chungcheong
  - Samsung Medical Center /ID# 248407, Seoul, Seoul Teugbyeolsi
- Taiwan (4):
  - Kaohsiung Chang Gung Memorial Hospital /ID# 248143, Kaohsiung City, Kaohsiung
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 248144, Kaohsiung City
  - National Cheng Kung University Hospital /ID# 248142, Tainan
  - Linkou Chang Gung Memorial Hospital /ID# 248145, Taoyuan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M22-137

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 9 participants were enrolled and received at least 1 dose of study drug.
Groups:
- Telisotuzumab Vedotin: Participants received telisotuzumab vedotin by intravenous (IV) infusion every 2 weeks until they met study drug discontinuation criteria.
Period: Overall Study
Arm/Group | Telisotuzumab Vedotin
Started | 9
Received at Least 1 Dose of Study Drug | 9
Completed | 0
Not Completed | 9
Not completed — Death | 4
Not completed — Study terminated by sponsor | 5

BASELINE CHARACTERISTICS:
Population: The efficacy evaluable analysis set included all participants who received at least 1 dose of study drug.
Groups:
- Telisotuzumab Vedotin: Participants received telisotuzumab vedotin by IV infusion every 2 weeks until they met study drug discontinuation criteria.
Arm/Group | Telisotuzumab Vedotin
Number analyzed (Participants) | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.4 (11.20)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 9
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) as Assessed by an Independent Central Review (ICR)
Description: ORR was defined as the percentage of participants with a confirmed complete response (CR) or confirmed partial response (PR) based on Response Evaluation Criteria in Solid Tumors (RECIST), version 1.1 as assessed by ICR.
Time Frame: Up to approximately 1.5 years
Population: The efficacy evaluable analysis set included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Telisotuzumab Vedotin
Number analyzed (Participants) | 9
percentage of participants | 33.3 [7.5 to 70.1]

2. Secondary Outcome: Duration of Response (DoR)
Description: DoR was defined for confirmed responders as the time from the initial response (CR or PR) to the first occurrence of radiographic progression per RECIST v1.1, or death from any cause.
Time Frame: Up to approximately 1.5 years
Population: The efficacy evaluable analysis set included all participants who received at least 1 dose of study drug. Here, "Overall number of participants analyzed" represents participants evaluable for this outcome measure with CR or PR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Telisotuzumab Vedotin
Number analyzed (Participants) | 3
months | 8.5 [2.5 to NA] — Not reached due to insufficient number of events.

3. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was defined as the percentage of participants with best overall response of confirmed CR or confirmed PR, or stable disease (SD) for at least 12 weeks following first dose of study drug, based on RECIST, version 1.1.
Time Frame: Up to approximately 1.5 years
Population: The efficacy evaluable analysis set included all participants who received at least 1 dose of study drug.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Telisotuzumab Vedotin
Number analyzed (Participants) | 9
percentage of participants | 44.4 [13.7 to 78.8]

4. Secondary Outcome: Progression Free Survival (PFS) Per ICR
Description: PFS was defined as the time from the participant's first dose of study drug to the first occurrence of radiographic progression based on RECIST, version 1.1 or death from any cause.
Time Frame: Up to approximately 1.5 years
Population: The efficacy evaluable analysis set included all participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Telisotuzumab Vedotin
Number analyzed (Participants) | 9
months | 4.0 [0.9 to NA] — Not reached due to insufficient number of events.

5. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time from participant's first dose of study drug to the event of death from any cause.
Time Frame: Up to approximately 1.5 years
Population: The efficacy evaluable analysis set included all participants who received at least 1 dose of study drug.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Telisotuzumab Vedotin
Number analyzed (Participants) | 9
months | 17.5 [0.9 to NA] — Not reached due to insufficient number of events.

6. Secondary Outcome: Change From Baseline in Cough as Measured by the Cough Item of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Lung Cancer Module 13 (EORTC QLQ-LC13)
Description: The cough item of the EORTC QLQ-LC13 was reported on a 0 to 100 scale, with higher scores representing worse health outcomes with increasing symptom levels or impacts. A negative change from baseline value indicated reduction (i.e. improvement) in symptoms.
Time Frame: Baseline, Day 1 of Cycles 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12, 13, 14, 15, 16, 17, 18, 19, 20, 21, 22, 23, 24, 25, 26, 28, 30, 32
Population: The efficacy evaluable analysis set included all participants who received at least 1 dose of study drug. Here, "Overall Number of Participants Analyzed" is the number of participants evaluable for this outcome measure, and "Number analyzed" is the number of participants evaluated at each time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telisotuzumab Vedotin
Number analyzed (Participants) | 8
score on a scale
  Cycle 2 Day 1 | -8.33 (15.430)
  Cycle 3 Day 1: number analyzed (Participants) | 6
  Cycle 3 Day 1 | -11.11 (34.427)
  Cycle 4 Day 1: number analyzed (Participants) | 6
  Cycle 4 Day 1 | -5.56 (13.608)
  Cycle 5 Day 1: number analyzed (Participants) | 6
  Cycle 5 Day 1 | -11.11 (17.213)
  Cycle 6 Day 1: number analyzed (Participants) | 5
  Cycle 6 Day 1 | -13.33 (29.814)
  Cycle 7 Day 1: number analyzed (Participants) | 5
  Cycle 7 Day 1 | -26.67 (27.889)
  Cycle 8 Day 1: number analyzed (Participants) | 4
  Cycle 8 Day 1 | -25.00 (31.914)
  Cycle 9 Day 1: number analyzed (Participants) | 5
  Cycle 9 Day 1 | -6.67 (14.907)
  Cycle 10 Day 1: number analyzed (Participants) | 5
  Cycle 10 Day 1 | -13.33 (18.257)
  Cycle 11 Day 1: number analyzed (Participants) | 4
  Cycle 11 Day 1 | -8.33 (16.667)
  Cycle 12 Day 1: number analyzed (Participants) | 2
  Cycle 12 Day 1 | -16.67 (23.570)
  Cycle 13 Day 1: number analyzed (Participants) | 2
  Cycle 13 Day 1 | -50.00 (23.570)
  Cycle 14 Day 1: number analyzed (Participants) | 1
  Cycle 14 Day 1 | -33.33 (NA) — SD not evaluable with n=1
  Cycle 15 Day 1: number analyzed (Participants) | 2
  Cycle 15 Day 1 | -16.67 (23.570)
  Cycle 16 Day 1: number analyzed (Participants) | 2
  Cycle 16 Day 1 | -33.33 (47.140)
  Cycle 17 Day 1: number analyzed (Participants) | 1
  Cycle 17 Day 1 | 0.00 (NA) — SD not evaluable with n=1
  Cycle 18 Day 1: number analyzed (Participants) | 1
  Cycle 18 Day 1 | 0.00 (NA) — SD not evaluable with n=1
  Cycle 19 Day 1: number analyzed (Participants) | 2
  Cycle 19 Day 1 | -50.00 (23.570)
  Cycle 20 Day 1: number analyzed (Participants) | 1
  Cycle 20 Day 1 | 0.00 (NA) — SD not evaluable with n=1
  Cycle 21 Day 1: number analyzed (Participants) | 1
  Cycle 21 Day 1 | -33.33 (NA) — SD not evaluable with n=1
  Cycle 22 Day 1: number analyzed (Participants) | 2
  Cycle 22 Day 1 | -50.00 (23.570)
  Cycle 23 Day 1: number analyzed (Participants) | 1
  Cycle 23 Day 1 | -33.33 (NA) — SD not evaluable with n=1
  Cycle 24 Day 1: number analyzed (Participants) | 1
  Cycle 24 Day 1 | -33.33 (NA) — SD not evaluable with n=1
  Cycle 25 Day 1: number analyzed (Participants) | 2
  Cycle 25 Day 1 | -50.00 (23.570)
  Cycle 26 Day 1: number analyzed (Participants) | 1
  Cycle 26 Day 1 | -33.33 (NA) — SD not evaluable with n=1
  Cycle 28 Day 1: number analyzed (Participants) | 2
  Cycle 28 Day 1 | -50.00 (23.570)
  Cycle 30 Day 1: number analyzed (Participants) | 1
  Cycle 30 Day 1 | -33.33 (NA) — SD not evaluable with n=1
  Cycle 32 Day 1: number analyzed (Participants) | 2
  Cycle 32 Day 1 | -33.33 (47.140)

7. Secondary Outcome: Change From Baseline in Pain as Measured by the Pain in Chest Item of the EORTC QLQ-LC13
Description: The pain in chest item of the EORTC QLQ-LC13 was reported on a 0 to 100 scale, with higher scores representing worse health outcomes with increasing symptom levels or impacts. A negative change from baseline value indicated reduction (i.e. improvement) in symptoms.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telisotuzumab Vedotin
Number analyzed (Participants) | 8
score on a scale
  Cycle 2 Day 1 | 4.17 (27.817)
  Cycle 3 Day 1: number analyzed (Participants) | 6
  Cycle 3 Day 1 | -5.56 (13.608)
  Cycle 4 Day 1: number analyzed (Participants) | 6
  Cycle 4 Day 1 | 5.56 (13.608)
  Cycle 5 Day 1: number analyzed (Participants) | 6
  Cycle 5 Day 1 | 16.67 (40.825)
  Cycle 6 Day 1: number analyzed (Participants) | 5
  Cycle 6 Day 1 | 0.00 (0.000)
  Cycle 7 Day 1: number analyzed (Participants) | 5
  Cycle 7 Day 1 | -6.67 (14.907)
  Cycle 8 Day 1: number analyzed (Participants) | 4
  Cycle 8 Day 1 | 0.00 (0.000)
  Cycle 9 Day 1: number analyzed (Participants) | 5
  Cycle 9 Day 1 | 0.00 (0.000)
  Cycle 10 Day 1: number analyzed (Participants) | 5
  Cycle 10 Day 1 | 0.00 (23.570)
  Cycle 11 Day 1: number analyzed (Participants) | 4
  Cycle 11 Day 1 | 8.33 (16.667)
  Cycle 12 Day 1: number analyzed (Participants) | 2
  Cycle 12 Day 1 | 0.00 (0.000)
  Cycle 13 Day 1: number analyzed (Participants) | 2
  Cycle 13 Day 1 | -16.67 (23.570)
  Cycle 14 Day 1: number analyzed (Participants) | 1
  Cycle 14 Day 1 | 0.00 (NA) — SD not evaluable with n=1
  Cycle 15 Day 1: number analyzed (Participants) | 2
  Cycle 15 Day 1 | 0.00 (0.000)
  Cycle 16 Day 1: number analyzed (Participants) | 2
  Cycle 16 Day 1 | 0.00 (0.000)
  Cycle 17 Day 1: number analyzed (Participants) | 1
  Cycle 17 Day 1 | 0.00 (NA) — SD not evaluable with n=1
  Cycle 18 Day 1: number analyzed (Participants) | 1
  Cycle 18 Day 1 | 0.00 (NA) — SD not evaluable with n=1
  Cycle 19 Day 1: number analyzed (Participants) | 2
  Cycle 19 Day 1 | 0.00 (0.000)
  Cycle 20 Day 1: number analyzed (Participants) | 1
  Cycle 20 Day 1 | 0.00 (NA) — SD not evaluable with n=1
  Cycle 21 Day 1: number analyzed (Participants) | 1
  Cycle 21 Day 1 | 0.00 (NA) — SD not evaluable with n=1
  Cycle 22 Day 1: number analyzed (Participants) | 2
  Cycle 22 Day 1 | 0.00 (0.000)
  Cycle 23 Day 1: number analyzed (Participants) | 1
  Cycle 23 Day 1 | 0.00 (NA) — SD not evaluable with n=1
  Cycle 24 Day 1: number analyzed (Participants) | 1
  Cycle 24 Day 1 | 0.00 (NA) — SD not evaluable with n=1
  Cycle 25 Day 1: number analyzed (Participants) | 2
  Cycle 25 Day 1 | -16.67 (23.570)
  Cycle 26 Day 1: number analyzed (Participants) | 1
  Cycle 26 Day 1 | 0.00 (NA) — SD not evaluable with n=1
  Cycle 28 Day 1: number analyzed (Participants) | 2
  Cycle 28 Day 1 | 0.00 (0.000)
  Cycle 30 Day 1: number analyzed (Participants) | 1
  Cycle 30 Day 1 | 0.00 (NA) — SD not evaluable with n=1
  Cycle 32 Day 1: number analyzed (Participants) | 2
  Cycle 32 Day 1 | 0.00 (0.000)

8. Secondary Outcome: Change From Baseline in Dyspnea as Measured by the Dyspnea Item of the EORTC QLQ-LC13
Description: The dyspnea item of the EORTC QLQ-LC13 was reported on a 0 to 100 scale, with higher scores representing worse health outcomes with increasing symptom levels or impacts. A negative change from baseline value indicated reduction (i.e. improvement) in symptoms.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telisotuzumab Vedotin
Number analyzed (Participants) | 8
score on a scale
  Cycle 2 Day 1 | -5.56 (16.798)
  Cycle 3 Day 1: number analyzed (Participants) | 6
  Cycle 3 Day 1 | -7.41 (11.476)
  Cycle 4 Day 1: number analyzed (Participants) | 6
  Cycle 4 Day 1 | 1.85 (4.536)
  Cycle 5 Day 1: number analyzed (Participants) | 6
  Cycle 5 Day 1 | 7.41 (9.072)
  Cycle 6 Day 1: number analyzed (Participants) | 5
  Cycle 6 Day 1 | 2.22 (4.969)
  Cycle 7 Day 1: number analyzed (Participants) | 5
  Cycle 7 Day 1 | -2.22 (12.172)
  Cycle 8 Day 1: number analyzed (Participants) | 4
  Cycle 8 Day 1 | -0.00 (9.072)
  Cycle 9 Day 1: number analyzed (Participants) | 5
  Cycle 9 Day 1 | 4.44 (6.086)
  Cycle 10 Day 1: number analyzed (Participants) | 5
  Cycle 10 Day 1 | -2.22 (12.172)
  Cycle 11 Day 1: number analyzed (Participants) | 4
  Cycle 11 Day 1 | -2.78 (13.981)
  Cycle 12 Day 1: number analyzed (Participants) | 2
  Cycle 12 Day 1 | 5.56 (7.857)
  Cycle 13 Day 1: number analyzed (Participants) | 2
  Cycle 13 Day 1 | -5.56 (23.570)
  Cycle 14 Day 1: number analyzed (Participants) | 1
  Cycle 14 Day 1 | 11.11 (NA) — SD not calculable with n=1
  Cycle 15 Day 1: number analyzed (Participants) | 2
  Cycle 15 Day 1 | 0.00 (0.000)
  Cycle 16 Day 1: number analyzed (Participants) | 2
  Cycle 16 Day 1 | -11.11 (15.713)
  Cycle 17 Day 1: number analyzed (Participants) | 1
  Cycle 17 Day 1 | 0.00 (NA) — SD not calculable with n=1
  Cycle 18 Day 1: number analyzed (Participants) | 1
  Cycle 18 Day 1 | 11.11 (NA) — SD not calculable with n=1
  Cycle 19 Day 1: number analyzed (Participants) | 2
  Cycle 19 Day 1 | -0.00 (15.713)
  Cycle 20 Day 1: number analyzed (Participants) | 1
  Cycle 20 Day 1 | 11.11 (NA) — SD not calculable with n=1
  Cycle 21 Day 1: number analyzed (Participants) | 1
  Cycle 21 Day 1 | 11.11 (NA) — SD not calculable with n=1
  Cycle 22 Day 1: number analyzed (Participants) | 2
  Cycle 22 Day 1 | -5.56 (23.570)
  Cycle 23 Day 1: number analyzed (Participants) | 1
  Cycle 23 Day 1 | 0.00 (NA) — SD not calculable with n=1
  Cycle 24 Day 1: number analyzed (Participants) | 1
  Cycle 24 Day 1 | 0.00 (NA) — SD not calculable with n=1
  Cycle 25 Day 1: number analyzed (Participants) | 2
  Cycle 25 Day 1 | 5.56 (7.857)
  Cycle 26 Day 1: number analyzed (Participants) | 1
  Cycle 26 Day 1 | 0.00 (NA) — SD not calculable with n=1
  Cycle 28 Day 1: number analyzed (Participants) | 2
  Cycle 28 Day 1 | -0.00 (15.713)
  Cycle 30 Day 1: number analyzed (Participants) | 1
  Cycle 30 Day 1 | 11.11 (NA) — SD not calculable with n=1
  Cycle 32 Day 1: number analyzed (Participants) | 2
  Cycle 32 Day 1 | -0.00 (15.713)

9. Secondary Outcome: Change From Baseline in Quality of Life as Measured by the Global Health Status/Quality of Life Domain of the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30).
Description: The Global Health Status/Quality of Life Domain of the EORTC QLQ-C30 was reported on a scale of 0 to 100, with higher scores indicating better global health status/functioning and a positive change from baseline indicating improvement.
Time Frame: as for outcome 6
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Telisotuzumab Vedotin
Number analyzed (Participants) | 8
score on a scale
  Cycle 2 Day 1 | 3.13 (14.042)
  Cycle 3 Day 1: number analyzed (Participants) | 6
  Cycle 3 Day 1 | 2.78 (12.546)
  Cycle 4 Day 1: number analyzed (Participants) | 6
  Cycle 4 Day 1 | -2.78 (8.607)
  Cycle 5 Day 1: number analyzed (Participants) | 6
  Cycle 5 Day 1 | -4.17 (14.672)
  Cycle 6 Day 1: number analyzed (Participants) | 5
  Cycle 6 Day 1 | 1.67 (12.360)
  Cycle 7 Day 1: number analyzed (Participants) | 5
  Cycle 7 Day 1 | 3.33 (7.454)
  Cycle 8 Day 1: number analyzed (Participants) | 4
  Cycle 8 Day 1 | 4.17 (8.333)
  Cycle 9 Day 1: number analyzed (Participants) | 5
  Cycle 9 Day 1 | -3.33 (18.257)
  Cycle 10 Day 1: number analyzed (Participants) | 5
  Cycle 10 Day 1 | 3.33 (7.454)
  Cycle 11 Day 1: number analyzed (Participants) | 4
  Cycle 11 Day 1 | -4.17 (8.333)
  Cycle 12 Day 1: number analyzed (Participants) | 2
  Cycle 12 Day 1 | 8.33 (11.785)
  Cycle 13 Day 1: number analyzed (Participants) | 2
  Cycle 13 Day 1 | 8.33 (11.785)
  Cycle 14 Day 1: number analyzed (Participants) | 1
  Cycle 14 Day 1 | 16.67 (NA) — SD not calculable with n=1
  Cycle 15 Day 1: number analyzed (Participants) | 2
  Cycle 15 Day 1 | 8.33 (11.785)
  Cycle 16 Day 1: number analyzed (Participants) | 2
  Cycle 16 Day 1 | 4.17 (5.893)
  Cycle 17 Day 1: number analyzed (Participants) | 1
  Cycle 17 Day 1 | 0.00 (NA) — SD not calculable with n=1
  Cycle 18 Day 1: number analyzed (Participants) | 1
  Cycle 18 Day 1 | 0.00 (NA) — SD not calculable with n=1
  Cycle 19 Day 1: number analyzed (Participants) | 2
  Cycle 19 Day 1 | -8.33 (11.785)
  Cycle 20 Day 1: number analyzed (Participants) | 1
  Cycle 20 Day 1 | 0.00 (NA) — SD not calculable with n=1
  Cycle 21 Day 1: number analyzed (Participants) | 1
  Cycle 21 Day 1 | 0.00 (NA) — SD not calculable with n=1
  Cycle 22 Day 1: number analyzed (Participants) | 2
  Cycle 22 Day 1 | -4.17 (5.893)
  Cycle 23 Day 1: number analyzed (Participants) | 1
  Cycle 23 Day 1 | -16.67 (NA) — SD not calculable with n=1
  Cycle 24 Day 1: number analyzed (Participants) | 1
  Cycle 24 Day 1 | 16.67 (NA) — SD not calculable with n=1
  Cycle 25 Day 1: number analyzed (Participants) | 2
  Cycle 25 Day 1 | 8.33 (11.785)
  Cycle 26 Day 1: number analyzed (Participants) | 1
  Cycle 26 Day 1 | 0.00 (NA) — SD not calculable with n=1
  Cycle 28 Day 1: number analyzed (Participants) | 2
  Cycle 28 Day 1 | -8.33 (11.785)
  Cycle 30 Day 1: number analyzed (Participants) | 1
  Cycle 30 Day 1 | 16.67 (NA) — SD not calculable with n=1
  Cycle 32 Day 1: number analyzed (Participants) | 2
  Cycle 32 Day 1 | -16.67 (23.570)

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the start of safety data collection (Day 1) to the end of the study. The median time on follow-up was 14.3 months.
Description: All-cause mortality and adverse events: all participants who received at least 1 dose of study drug.
Arm/Group | Telisotuzumab Vedotin
All-Cause Mortality (participants affected / at risk) | 4/9
Serious Adverse Events (participants affected / at risk) | 3/9
Other Adverse Events (participants affected / at risk) | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telisotuzumab Vedotin (N=9)
DIARRHOEA (Gastrointestinal disorders) | 1 (1)
INTESTINAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
DISEASE PROGRESSION (General disorders) | 2 (2)
PNEUMONIA (Infections and infestations) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Telisotuzumab Vedotin (N=9)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1)
KERATITIS (Eye disorders) | 2 (4)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 3 (3)
ASTHENIA (General disorders) | 3 (3)
DISEASE PROGRESSION (General disorders) | 1 (1)
FATIGUE (General disorders) | 2 (3)
MEDICAL DEVICE PAIN (General disorders) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 2 (2)
PYREXIA (General disorders) | 1 (1)
CHOLESTASIS (Hepatobiliary disorders) | 1 (1)
ORAL FUNGAL INFECTION (Infections and infestations) | 1 (1)
LIGAMENT SPRAIN (Injury, poisoning and procedural complications) | 1 (1)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 2 (2)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 1 (1)
BLOOD GLUCOSE INCREASED (Investigations) | 1 (1)
BLOOD TESTOSTERONE DECREASED (Investigations) | 1 (1)
C-REACTIVE PROTEIN INCREASED (Investigations) | 1 (1)
LYMPHOCYTE COUNT DECREASED (Investigations) | 1 (2)
NEUTROPHIL COUNT INCREASED (Investigations) | 1 (1)
WEIGHT DECREASED (Investigations) | 1 (1)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 1 (2)
DECREASED APPETITE (Metabolism and nutrition disorders) | 1 (1)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 2 (2)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 1 (2)
PRESYNCOPE (Nervous system disorders) | 1 (1)
TASTE DISORDER (Nervous system disorders) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HAEMOPTYSIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PULMONARY HAEMORRHAGE (Respiratory, thoracic and mediastinal disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (3)
RASH (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2023-03-07): https://cdn.clinicaltrials.gov/large-docs/03/NCT05513703/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT05513703/SAP_001.pdf